CLINICAL TRIAL: NCT04415983
Title: Study of Novel Triple Nitazoxanide (NTZ) Based New Therapeutic Regimens for Helicobacter Pylori in Children
Brief Title: Study of Nitazoxanide (NTZ) for Helicobacter Pylori in Children
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: helicobacter children
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — nitazoxanide; Clarithromycin; Metronidazole; Proton Pump Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide group (Experimental): Clarithromycin, Nitazoxanide and Proton pump inhibitor
  Interventions: Drug: Nitazoxanide; Drug: Clarithromycin; Drug: Proton pump inhibitor
- Traditional group (Active Comparator): Clarithromycin, Metronidazole and Proton pump inhibitor
  Interventions: Drug: Clarithromycin; Drug: Metronidazole; Drug: Proton pump inhibitor

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide twice daily
  Other Names: nanazoxid
  Arms: Nitazoxanide group
Drug: Clarithromycin — Klacid twice daily
  Other Names: Klacid
Drug: Metronidazole — Metronidazole twice daily
  Other Names: Flagyl
  Arms: Traditional group
Drug: Proton pump inhibitor — Omeprazoe twice daily

SUMMARY:
Study of Nitazoxanide (NTZ) based therapeutic regimens for Helicobacter pylori in children

DETAILED DESCRIPTION:
Study of Novel triple Nitazoxanide (NTZ) based new therapeutic regimens for Helicobacter pylori in children

ELIGIBILITY:
Inclusion Criteria:

- Positive helicobacter infection.

Exclusion Criteria:

* Previous treatment for H. Pylori.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with cured helicobacter infection | 6 months
  Total number of patients with eradicated helicobacter infection

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Gamal, Ass. Prof., Principal Investigator — Pediatrics department - Tanta University; sherief Abd-Elsalam, ass. Prof., Principal Investigator — Tanta University Faculty of medicine; Abeer Salamah, Lecturer, Study Director — Pediatrics department - Kafr Elsheikh University; dina shawky, lecturer, Study Director — Pediatrics department - Tanta University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No